CLINICAL TRIAL: NCT04017286
Title: A Prospective Cohort Study of the Association Between Pregnancy Health and Offspring Developmental & Behavioral Outcomes(Multi-Centered)
Brief Title: Relationship About Pregnancy Health and Offspring Developmental &Behavioral Outcomes
Acronym: APCSAHAODBO
Status: Recruiting | Type: Observational
Sponsor: Chen Li (Other)
Responsible Party: Sponsor-Investigator, Chen Li, Vice Director, Professor, Children's Hospital of Chongqing Medical University
Organization: Children's Hospital of Chongqing Medical University (Other)
Other Study IDs: CLi
Record Dates: First submitted 2018-05-21; First posted 2019-07-12 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Children Behavior Problem; Pregnancy
Keywords: Developmental assessment; Homocysteine; physique growth; nutrients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Biospecimen Retention: Samples With DNA — In the investigator's study, partly samples of material from research participants are retained in a biorepository.For example, cord blood from newborn, DNA, venous blood and urine. A few of hair is also collected at the same time and stored for future measurements (used to extract DNA in case that the cord blood is unsufficient or DNA extraction from the blood fails unexpectedly).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (4):
- depressive disorder group: At 21 weeks of pregnancy, women diagnosed with depressive disorder by the Hamilton depression scale and Beck depression rating scale and their offspring were enrolled.
- Nutrient-deficient group: Nutrients (Vitamin A,D,E) were tested at 21 weeks of pregnancy, and pregnant women with one or more nutrient deficiencies or insufficiency and their offspring were enrolled.
- depressive disorder and nutrient deficiency group: At 21 weeks of pregnancy, pregnant women with depressive disorder and nutrient deficiency or insufficiency and their offspring were enrolled.
- Neither group: At 21 weeks of pregnancy, pregnant women without depressive disorder and nutrient deficiency or insufficiency and their offspring were enrolled.

SUMMARY:
This topic puts forward a hypothesis: genetic and environmental factors such as major depressive disorder during pregnancy, nutritional status of vitamin A, D, E, and folic acid, intestinal microecology, and bisphenol A exposure, may affect the cognitive development level of the offspring through the genetic correlation with attention deficit hyperactivity disorder, developmental delay/intellectual disability, and major depressive disorder, allelic heterogeneity and pleiotropy of ITIH3 mediated by SNP and CACNB2, neurotransmitters like dopamine, and metabolic pathways, thereby increasing the risk of attention deficit hyperactivity disorder and developmental delay/intellectual disability prevalence on offspring.

This topic planning from allelic heterogeneity and pleiotropy of attention deficit hyperactivity disorder and major depressive disorder mediated by SNP, neurotransmitters like dopamine, and metabolic pathways, explores deeply the influences on children's development level and the risk of common neurological disorder caused by genetic and environmental factors during pregnancy, looking for reasonable prevention, early diagnosis of biomarkers and therapeutic targets, in order to provide data support for further improvement and revision of national mother and infant healthcare policy .

DETAILED DESCRIPTION:
1. Technology Roadmap:①Pregnant Women:Subjects are rolled in the group. ② 21 Weeks of Gestation：Sign informed contents (mother version), test depression scale ( BDI+HAMD ), fill in the basic information questionnaire and collect 3 ml of blood of pregnant women for genetic information extraction. ③Delivery: Sign informed contents(children version), collect 1 ml of umbilical cord blood and 2ml of urine from mother. ④Physical measurements are respectively taken when a child is 3, 6, 12, 24 months old and 3, 6 years old. And the Montreal Children Hospital Feeding Scale will be also respectively completed when a child is 6 and 12 months old. What's more, the investigators plan to carry out developmental screening for the children aged 1, 2, 3 and 6, and if the developmental screening is positive, a diagnostic test then will be carried out. ⑤When children are aged 2, 3 and 6, blood samples are taken from 3 milliliters and urine from 2 milliliters, and nutrients are detected to obtain genetic information. ⑥All biological specimens will be tested for nutrient levels and some other.⑦At last, data analysis is performed on all collected information including physical measurements, feeding behavior questionnaire, all biological specimens and so on.
2. Study Protocol： A. Human Subjects Review: Studies must have approval (or be exempt, as appropriate) from a Human Subjects Protection Review Board prior to the enrollment of the first participant to be eligible for registration (Submitted, approved).

   B. Register a clinical study: Prior to the launch of the project, pre-registration will be completed at clinicaltrials.gov in the international clinical study register authority.

   C. Study cohort: Screening qualified pregnant women volunteered to take part in the study from pregnancy clinics of Chongqing suburban maternity and child health hospital and The Maternal and Child Health Hospital of Hainan Province.
3. Measuring scale: To assess the depression status and degree of the subjects by Hamilton Depression Scale (HAMD) and Beck depression rating scale (BDI); To evaluate the cognitive function of subjects and exclude the patients with mental retardation by Mini-Mental State Examination (MMSE) and Activity of Daily Living Scale（ADL); To screen or identify the cognitive function and level of children in different age groups by Denver development screening scale (DDST) and Gesell Developmental Schedules (Gesell), and combining with the Adaptive Scale of Infant and Children (SM) to assist in the diagnosis of developmental delay/intellectual disability, The Vanderbilt ADHD Diagnostic Rating Scale on diagnosis of ADHD.
4. Data management and statistical analysis plan:

   A. All the data is recorded by the professional staff, and checked by a third person to ensure accuracy of data entry; B. All statistical analysis is performed with SAS 9.4. The statistical analysis is completed by the applicant and the professional statisticians in the epidemiology research office of the unit.
5. Recruitment process:

   A. To preach related knowledge of major depressive disorder, ADHD, and developmental delay/intellectual disability in the form of obstetrics clinics, network media, and network health management platform,etc; B. Recruitment information is released by platforms such as obstetrics clinics, network health management platforms, etc., to recruit pregnant women; C. The obstetric nurses and professional recruiters (postgraduate students) assist pregnant women to sign informed consents, agree to participate in the study, and promise that the delivery of children would take part in the same sequence of study as well.
6. The required materials of recruitment:

   Manufacture recruiting advertisements of major depressive disorder, ADHD, developmental delay/intellectual disability related knowledge and disease hazards, the importance of early diagnosis, recruitment information of pregnant women and their children enrolled in the study (for example: network media recruitment advertisement, WeChat H5 recruitment advertisement, network health management platform recruitment advertisement, etc.).
7. Benefit Assessment： A. The pregnant women volunteered to participate in the study are able to enjoy regular check-ups (once every three months, including height, weight, blood pressure, mood questionnaires, etc.); B. Eligible children volunteer to participate in the study, all can enjoy free physical examination (height, weight) at the age of 1, 2, 3, and 6, moreover according to age to enjoy free screening or diagnostic test related to cognitive development level and attention deficit hyperactivity disorder test; C. The parents of all the children involved can receive the knowledge of parenting through WeChat or network health management platform, and be provided with free parenting seminars regularly; D. High-risk pregnant women and children are given priority access to the superior hospital for diagnosis and treatment; E. All subjects are eligible for the the nutrient level test of preferential price, 16S test (intestinal flora detection) of the preferential price , free related genetic test; F. Study may solve some urgent problems in the prevention and treatment of developmental disabilities such as ADHD, developmental delay/intellectual disability, and contribute to promoting maternal and child health, improving the quality of the population, and promoting the sustained and healthy development of the national economy.
8. Risk Assessment ( illustrate the possible risk rate and take measures to ensure that risk is minimized in a possible range):

   A. Possible risk: the probability of subjects losing to follow-up (loss ratio of 5 to 10% due to various reasons); B. Measurements: The professional staff would regularly contact with the mother or the child by phone or Wechat. And after the birth of a child, childbearing knowledge or childcare lectures are regularly provided for the parents.
9. Special crowd protection:

A.In the course of the study, obstetricians, psychologists, and childcare doctors are all involved in providing health care for pregnant women, mothers and children.

B. At the same time, please protect the subjects' privacy and not to give out the information of the subjects. All subjects' personal information is treated with confidentiality and this study data is only used in the study design scope to ensure that the subjects' privacy is not invaded.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion criteria for pregnant women: Aged 20~49;
2. no cognitive impairment, able to complete the scale test;
3. Hamilton Depression Scale (HAMD questionnaire) is normal (HAMD score <8 points) or mild to moderate positive (HAMD questionnaire score: 8~35 points);
4. Participants are asked for their own written informed content for the study;

Exclusion Criteria:

1. Patients receiving anti-depression therapy during the first 6 months of gestation or during pregnancy;
2. Patients with severe depression with scores of no less than 35 points in the HAMD questionnaire;
3. Patients with other mental disorders;
4. Patients with neurological diseases;
5. Patients with cognitive dysfunction.

Ages: 3 Months to 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study is based on source material from Chongqing suburban maternity and child health hospital. The investigators randomly select the pregnant women aged 20 to 49 from the pregnancy clinics and obstetric wards, respectively construct mother-child matching and a prospective study cohort depending on whether the pregnant women with major depressive disorder or not, nutrition state of vitamin A, D, E, during pregnancy.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Denver Developmental Screening Test results within 72 months of age | 72 months
  The DDST is taking at the age of 12 months,24 months,36months and 72months respectively ,consists of 104 items, spread 4 domains, such as gross motor, fine motor, language and personal-social skill. A normal score means no delay in any domain and no more than one caution; an abnormal score means two or more domains with two or more delays or one domain with two or more delays and another domains with one delay; a suspect score means one or more domains with one delay and more than one cautions or one domain with two or more delays; a score of untestable means enough refused items that the score would be suspect if they had been delays.
Changes in Gesell Developmental Schedules test results within 72 months of age | 72 months
  The GDS is taking at the age of 12 months,24 months, 36 months and 72 months respectively , evaluate a child's cognitive, language, motor and social-emotional responses in five strands: adaptation, gross motor, fine motor, language and personal-social skill, then schedule operates off what is known as an individual's developmental quotient (DQ). Diagnostic criteria: the score of DQ≥86: normal, 76-85: marginal , 55-75: mild mental retardation, 40-54: moderate mental retardation, 25-39: severe mental retardation, and ≤25 : extremely severe mental retardation.
The Vanderbilt Attention Deficit Hyperactivity Disorder Diagnostic Rating Scale | 72 months
  The Vanderbilt ADHD Diagnostic Rating Scale (VADRS) is for children at the age of 72 months. Scores of 2 or 3 on a single Symptom question reflect often-occurring behaviors. Scores of 4 or 5 on Performance questions reflect problems in performance. To meet the diagnosis of ADHD, one must have at least 6 positive responses to either the inattentive 9 or hyperactive 9 core symptoms, or both.
Changes in vitamin A | 72 months
  Vitamin A is measured for the mothers at first visit during 21 weeks of gestation and delivery, for the children is 24 months, 36 months and 72 months respectively. It is measured by HPLC and tandem mass spectrometry. And it is considered as Vitamin A deficiency when the concentration is below 0.70 umol/L, 0.70-1.05 umol/L is considered as marginal vitamin A deficiency, 1.05-2.56 umol/L is considered as normal range, and over 2.56 umol/L is considered as Vitamin A excess.
Changes in Vitamin D | 72 months
  Vitamin D is measured for the mothers at first visit during 21 weeks of gestation and delivery, for the children is 24 months, 36 months and 72 months respectively. It is measured by HPLC and tandem mass spectrometry. the measurement of the concentration of 25-OH-D3 as that of vitamin D. It is below 30 nmol/L considered as Vitamin D deficiency, 30-50 nmol/L considered as Vitamin D insufficiency, over 50 nmol/L considered as Vitamin D sufficiency.
Changes in Vitamin E | 72 months
  Vitamin E is measured for the mothers at first visit during 21 weeks of gestation and delivery, for the children is 24 months, 36 months and 72 months respectively. It is measured by HPLC and tandem mass spectrometry. It is normal range with the concentration of 11.6-46.4 umol/L.
Homocysteine | delivery
  Homocysteine is measured for the mothers at first visit during 21 weeks of gestation and delivery. It is measured by HPLC and tandem mass spectrometry. The concentration of homocysteine less than 11.4umol/L is normal for men and less than 10.4 umol/L for women.
Bisphenol A | 72 months
  The concentration of bisphenol A is measured for mother at delivery and for children aged 2 and 6. The investigators measured the concentration of urine in order to compare the differences of children between high dose of BPA with low dose of BPA. However, as far as we know, the normal range of bisphenol A has not been reported at home and abroad. We also want to explore the relationship between bisphenol A and neuropsychiatric development.
the Adaptive Scale of Infant and Children | 72 months
  This scale is assessed for the children at the age of 72 months. Extremely low (≤5), severely low (6 points), moderately low (8 points), marginal (9 points), normal (10 points), more than normal (11 points), excellent (12 points), very good (13 points).

SECONDARY OUTCOMES:
Beck depression rating scale | 21 weeks of pregnancy
  The investigators assess Beck depression rating scale the severity of depression of the women at 21 weeks of pregnancy by Beck depression rating scale, a 21-items questionnaire. Scoring criteria: 0-13: good mental state, 14-19: mildly depressed, 20-28: moderately depressed, 29-63: severe depression.
Hamilton Depression Scale | 21 weeks of pregnancy
  The investigators assess the mood of the pregnant women at 21 weeks of pregnancy by the scale. Total score < 8: normal; A score of 8 to 20: possible depression; A score of 20 to 35: depression; Overall score > 35: major depression.
Mini-Mental State Examination | 21 weeks of pregnancy
  The investigators screened the questionnaire to assess cognitive impairment of the pregnant women at 21 weeks of pregnancy. Any score greater than or equal to 24 points (out of 30) indicates a normal cognition. Below this, scores can indicate severe (≤9 points), moderate (10-18 points) or mild (19-23 points) cognitive impairment.
Changes in the Montreal Children Hospital Feeding Scale within 12 months of age | 12 months
  The scale measured for the children aged 6 months and 12 months respectively. The score previously calculated is the original score without standardization (rough score), and the total score of the scale (rough score) is 14-98, and then the rough score is converted into standardized score. If the standard score is less than or equal to 50, there is no difficulty in feeding; if the standard score is 51-60, there is mild difficulty in feeding; if the standard score is 61-70, there is moderate difficulty in feeding; if the standard score is greater than 70, there is severe difficulty in feeding.
Change of weight for height Z-score(WHZ) | 72 months
  The measurement of body length/height and weight (the average of three consecutive measurements) for age is at 3 months, 6 months,12 months,24 months,36 months and 72 months respectively and calculated by WHO2006 curve. It's considered abnormal when the WHZ is below P3 or over P97, the normal range is between P3~P97.
Change of the height for age Z-score(HAZ) | 72 months
  The measurement of body length/height (the average of three consecutive measurements) for age is at 3 months, 6 months,12 months , 24 months, 36 months and 72 months respectively and calculated by WHO2006 curve. It's considered abnormal when the HAZ is below P3 or over P97, the normal range is between P3~P97.
Change of the weight for Age Z-score(WAZ) | 72 months
  The measurement of weight (the average of three consecutive measurements) for age is at 3 months, 6 months,12 months , 24 months, 36 months and 72 months respectively and calculated by WHO2006 curve . It's considered abnormal when the WAZ is below P3 or over P97, the normal range is between P3~P97.
Ferritin | 24 months
  The ferritin is measured for mothers at 21 weeks of pregnancy and for children at the age of 24 months. It is measured by chemiluminescence method. It is normal when the concentration of ferritin is between 5-148 ng/ml for girls and 28-365 ng/ml for boys.
Folate | 24 months
  The folate is measured for mothers at 21 weeks of pregnancy and for children at the age of 24 months. It is measured by chemiluminescence method. It is normal when the concentration of folate is greater than 5.38 ng/ml.
Activity of Daily Living Scale | 21 weeks of pregnancy
  The investigators screened the questionnaire to assess cognitive impairment of the pregnant women at 21 weeks of pregnancy. ADLs can be broken down into the following categories: personal hygiene, continence management, dressing, feeding, ambulating. The evaluation results can be analyzed according to the total score, subscale score and single score. The total score < 16 points, completely normal; > 16 points, with varying degrees of functional decline, and the maximum score is 64 points. Single points; 1 point :normal, 2-4 points : functional decline.≥2 items with a score ≥3 points, or a total score ≥ 22 points, are considered to have obvious dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Li Chen, MD, Study Director — Children's Hospital of Chongqing Medical University; Tanya Froehlich, MD,MS, Principal Investigator — Children's Hospital Medical Center, Cincinnati; yu T Li, MS, Study Chair — Children's Hospital of Chongqing Medical University
Locations (5):
- China (5):
  - The People's Hospital of Yubei District of Chongqing City, Chongqing, Chongqing Municipality
  - Chongqing First People's Hospital of Liangjiang New Area, Chongqing, Chongqing Municipality
  - The Central Hospital of Jiangjin District of Chongqing City, Chongqing, Chongqing Municipality
  - Wanzhou Health Center for Women and Children, Chongqing, Chongqing Municipality
  - The Maternal and Child Health Hospital of Hainan Province, Haikou, Hainan

IPD SHARING:
Plan to Share IPD: No
Data is confidential during the study.

REFERENCES:
- [Background] Zeng J, Chen L, Wang Z, Chen Q, Fan Z, Jiang H, Wu Y, Ren L, Chen J, Li T, Song W. Marginal vitamin A deficiency facilitates Alzheimer's pathogenesis. Acta Neuropathol. 2017 Jun;133(6):967-982. doi: 10.1007/s00401-017-1669-y. Epub 2017 Jan 27. PMID 28130638
- [Background] Zeng J, Li T, Gong M, Jiang W, Yang T, Chen J, Liu Y, Chen L. Marginal Vitamin A Deficiency Exacerbates Memory Deficits Following Abeta1-42 Injection in Rats. Curr Alzheimer Res. 2017;14(5):562-570. doi: 10.2174/1567205013666161223162110. PMID 28017127
- [Background] Liu Y, Chen Q, Wei X, Chen L, Zhang X, Chen K, Chen J, Li T. Relationship between perinatal antioxidant vitamin and heavy metal levels and the growth and cognitive development of children at 5 years of age. Asia Pac J Clin Nutr. 2015;24(4):650-8. doi: 10.6133/apjcn.2015.24.4.25. PMID 26693750
- [Background] Hanson C, Lyden E, Furtado J, Van Ormer M, Schumacher M, Kamil A, McGinn E, Rilett K, Elliott E, Cave C, Johnson R, Weishaar K, Anderson-Berry A. Vitamin E status and associations in maternal-infant Dyads in the Midwestern United States. Clin Nutr. 2019 Apr;38(2):934-939. doi: 10.1016/j.clnu.2018.02.003. Epub 2018 Feb 20. PMID 29496275
- [Background] Biederman J, Faraone SV. Attention-deficit hyperactivity disorder. Lancet. 2005 Jul 16-22;366(9481):237-48. doi: 10.1016/S0140-6736(05)66915-2. PMID 16023516
- [Background] Barker DJ, Osmond C. Infant mortality, childhood nutrition, and ischaemic heart disease in England and Wales. Lancet. 1986 May 10;1(8489):1077-81. doi: 10.1016/s0140-6736(86)91340-1. PMID 2871345
- [Background] Lin Y, Xu J, Huang J, Jia Y, Zhang J, Yan C, Zhang J. Effects of prenatal and postnatal maternal emotional stress on toddlers' cognitive and temperamental development. J Affect Disord. 2017 Jan 1;207:9-17. doi: 10.1016/j.jad.2016.09.010. Epub 2016 Sep 19. PMID 27665073
- [Background] Ferguson SS. Receptor tyrosine kinase transactivation: fine-tuning synaptic transmission. Trends Neurosci. 2003 Mar;26(3):119-22. doi: 10.1016/S0166-2236(03)00022-5. PMID 12591212
- [Background] Vinkhuyzen AAE, Eyles DW, Burne THJ, Blanken LME, Kruithof CJ, Verhulst F, Jaddoe VW, Tiemeier H, McGrath JJ. Gestational vitamin D deficiency and autism-related traits: the Generation R Study. Mol Psychiatry. 2018 Feb;23(2):240-246. doi: 10.1038/mp.2016.213. Epub 2016 Nov 29. PMID 27895322
- [Background] Salucci S, Ambrogini P, Lattanzi D, Betti M, Gobbi P, Galati C, Galli F, Cuppini R, Minelli A. Maternal dietary loads of alpha-tocopherol increase synapse density and glial synaptic coverage in the hippocampus of adult offspring. Eur J Histochem. 2014 May 2;58(2):2355. doi: 10.4081/ejh.2014.2355. PMID 24998923
- [Background] Hanson M. The birth and future health of DOHaD. J Dev Orig Health Dis. 2015 Oct;6(5):434-7. doi: 10.1017/S2040174415001129. Epub 2015 May 25. PMID 26004094
- [Background] Zhao H, Nyholt DR. Gene-based analyses reveal novel genetic overlap and allelic heterogeneity across five major psychiatric disorders. Hum Genet. 2017 Feb;136(2):263-274. doi: 10.1007/s00439-016-1755-6. Epub 2016 Dec 29. PMID 28035465
- [Background] Dias CC, Figueiredo B, Pinto TM. Children's Sleep Habits Questionnaire - Infant Version. J Pediatr (Rio J). 2018 Mar-Apr;94(2):146-154. doi: 10.1016/j.jped.2017.05.012. Epub 2017 Aug 23. PMID 28842258
- [Background] Cross-Disorder Group of the Psychiatric Genomics Consortium; Lee SH, Ripke S, Neale BM, Faraone SV, Purcell SM, Perlis RH, Mowry BJ, Thapar A, Goddard ME, Witte JS, Absher D, Agartz I, Akil H, Amin F, Andreassen OA, Anjorin A, Anney R, Anttila V, Arking DE, Asherson P, Azevedo MH, Backlund L, Badner JA, Bailey AJ, Banaschewski T, Barchas JD, Barnes MR, Barrett TB, Bass N, Battaglia A, Bauer M, Bayes M, Bellivier F, Bergen SE, Berrettini W, Betancur C, Bettecken T, Biederman J, Binder EB, Black DW, Blackwood DH, Bloss CS, Boehnke M, Boomsma DI, Breen G, Breuer R, Bruggeman R, Cormican P, Buccola NG, Buitelaar JK, Bunney WE, Buxbaum JD, Byerley WF, Byrne EM, Caesar S, Cahn W, Cantor RM, Casas M, Chakravarti A, Chambert K, Choudhury K, Cichon S, Cloninger CR, Collier DA, Cook EH, Coon H, Cormand B, Corvin A, Coryell WH, Craig DW, Craig IW, Crosbie J, Cuccaro ML, Curtis D, Czamara D, Datta S, Dawson G, Day R, De Geus EJ, Degenhardt F, Djurovic S, Donohoe GJ, Doyle AE, Duan J, Dudbridge F, Duketis E, Ebstein RP, Edenberg HJ, Elia J, Ennis S, Etain B, Fanous A, Farmer AE, Ferrier IN, Flickinger M, Fombonne E, Foroud T, Frank J, Franke B, Fraser C, Freedman R, Freimer NB, Freitag CM, Friedl M, Frisen L, Gallagher L, Gejman PV, Georgieva L, Gershon ES, Geschwind DH, Giegling I, Gill M, Gordon SD, Gordon-Smith K, Green EK, Greenwood TA, Grice DE, Gross M, Grozeva D, Guan W, Gurling H, De Haan L, Haines JL, Hakonarson H, Hallmayer J, Hamilton SP, Hamshere ML, Hansen TF, Hartmann AM, Hautzinger M, Heath AC, Henders AK, Herms S, Hickie IB, Hipolito M, Hoefels S, Holmans PA, Holsboer F, Hoogendijk WJ, Hottenga JJ, Hultman CM, Hus V, Ingason A, Ising M, Jamain S, Jones EG, Jones I, Jones L, Tzeng JY, Kahler AK, Kahn RS, Kandaswamy R, Keller MC, Kennedy JL, Kenny E, Kent L, Kim Y, Kirov GK, Klauck SM, Klei L, Knowles JA, Kohli MA, Koller DL, Konte B, Korszun A, Krabbendam L, Krasucki R, Kuntsi J, Kwan P, Landen M, Langstrom N, Lathrop M, Lawrence J, Lawson WB, Leboyer M, Ledbetter DH, Lee PH, Lencz T, Lesch KP, Levinson DF, Lewis CM, Li J, Lichtenstein P, Lieberman JA, Lin DY, Linszen DH, Liu C, Lohoff FW, Loo SK, Lord C, Lowe JK, Lucae S, MacIntyre DJ, Madden PA, Maestrini E, Magnusson PK, Mahon PB, Maier W, Malhotra AK, Mane SM, Martin CL, Martin NG, Mattheisen M, Matthews K, Mattingsdal M, McCarroll SA, McGhee KA, McGough JJ, McGrath PJ, McGuffin P, McInnis MG, McIntosh A, McKinney R, McLean AW, McMahon FJ, McMahon WM, McQuillin A, Medeiros H, Medland SE, Meier S, Melle I, Meng F, Meyer J, Middeldorp CM, Middleton L, Milanova V, Miranda A, Monaco AP, Montgomery GW, Moran JL, Moreno-De-Luca D, Morken G, Morris DW, Morrow EM, Moskvina V, Muglia P, Muhleisen TW, Muir WJ, Muller-Myhsok B, Murtha M, Myers RM, Myin-Germeys I, Neale MC, Nelson SF, Nievergelt CM, Nikolov I, Nimgaonkar V, Nolen WA, Nothen MM, Nurnberger JI, Nwulia EA, Nyholt DR, O'Dushlaine C, Oades RD, Olincy A, Oliveira G, Olsen L, Ophoff RA, Osby U, Owen MJ, Palotie A, Parr JR, Paterson AD, Pato CN, Pato MT, Penninx BW, Pergadia ML, Pericak-Vance MA, Pickard BS, Pimm J, Piven J, Posthuma D, Potash JB, Poustka F, Propping P, Puri V, Quested DJ, Quinn EM, Ramos-Quiroga JA, Rasmussen HB, Raychaudhuri S, Rehnstrom K, Reif A, Ribases M, Rice JP, Rietschel M, Roeder K, Roeyers H, Rossin L, Rothenberger A, Rouleau G, Ruderfer D, Rujescu D, Sanders AR, Sanders SJ, Santangelo SL, Sergeant JA, Schachar R, Schalling M, Schatzberg AF, Scheftner WA, Schellenberg GD, Scherer SW, Schork NJ, Schulze TG, Schumacher J, Schwarz M, Scolnick E, Scott LJ, Shi J, Shilling PD, Shyn SI, Silverman JM, Slager SL, Smalley SL, Smit JH, Smith EN, Sonuga-Barke EJ, St Clair D, State M, Steffens M, Steinhausen HC, Strauss JS, Strohmaier J, Stroup TS, Sutcliffe JS, Szatmari P, Szelinger S, Thirumalai S, Thompson RC, Todorov AA, Tozzi F, Treutlein J, Uhr M, van den Oord EJ, Van Grootheest G, Van Os J, Vicente AM, Vieland VJ, Vincent JB, Visscher PM, Walsh CA, Wassink TH, Watson SJ, Weissman MM, Werge T, Wienker TF, Wijsman EM, Willemsen G, Williams N, Willsey AJ, Witt SH, Xu W, Young AH, Yu TW, Zammit S, Zandi PP, Zhang P, Zitman FG, Zollner S, Devlin B, Kelsoe JR, Sklar P, Daly MJ, O'Donovan MC, Craddock N, Sullivan PF, Smoller JW, Kendler KS, Wray NR; International Inflammatory Bowel Disease Genetics Consortium (IIBDGC). Genetic relationship between five psychiatric disorders estimated from genome-wide SNPs. Nat Genet. 2013 Sep;45(9):984-94. doi: 10.1038/ng.2711. Epub 2013 Aug 11. PMID 23933821
- [Derived] Zhao W, Li C, Shen WZ, Li KY, Cai YX, Li F, Fu H, Peng B, Chen J, Li TY, Chen L. Cord blood vitamin A and vitamin D levels in relation to physical growth in exclusively breastfed infants aged 0-6 months. Front Endocrinol (Lausanne). 2024 Jul 26;15:1394408. doi: 10.3389/fendo.2024.1394408. eCollection 2024. PMID 39129921